CLINICAL TRIAL: NCT02058550
Title: Phase I Pilot Study Evaluating Vaginal Dilator Use and Toxicity Following Vaginal Brachytherapy
Brief Title: Phone or Email Reminder in Increasing Vaginal Dilator Use in Patients With Gynecologic Cancers Undergoing Brachytherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-29074; NCI-2013-02400 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GYN0005 (Other: OnCore)
Record Dates: First submitted 2014-02-06; First posted 2014-02-10 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Cervical Cancer; Endometrial Cancer; Radiation Toxicity; Vaginal Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Radiation Injuries; Vaginal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm I (no intervention) (No Intervention): Patients receive no additional reminders.
- Arm II (email survey) (Experimental): Patients receive a reminder email survey every 2 weeks for 1 year after completing radiation.
  Interventions: Other: survey administration; Other: computer-assisted intervention
- Arm III (email surveys and phone calls) (Experimental): Patients receive a reminder email survey as in Arm I and 4 additional phone calls at 4-8 weeks, 3-5 months, 7-8 months, and 10-11 months during their first year of follow-up.
  Interventions: Other: survey administration; Other: computer-assisted intervention; Behavioral: telephone-based intervention

INTERVENTIONS:
Other: survey administration — Receive reminder email survey
  Arms: Arm II (email survey); Arm III (email surveys and phone calls)
Other: computer-assisted intervention — Receive reminder email survey
  Arms: Arm II (email survey); Arm III (email surveys and phone calls)
Behavioral: telephone-based intervention — Receive reminder phone call
  Arms: Arm III (email surveys and phone calls)

SUMMARY:
This randomized, pilot phase I trial studies whether phone or email reminders increases vaginal dilator use in patients with endometrial, cervical, or vaginal cancers after they undergo brachytherapy. Brachytherapy is a type of internal radiation which uses radioactive material placed directly into or near a tumor to kill tumor cells. A reminder program may help increase use of vaginal dilators and decrease long-term side effects following brachytherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate whether vaginal dilator adherence is improved with additional reminder phone calls and/or email reminder survey.

SECONDARY OBJECTIVES:

I. Evaluate whether there are differences in the length of vaginal canal between the non-intervention and intervention groups. Evaluate rates of gynecologic, urinary, and gastrointestinal toxicity.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM I: Patients receive no additional reminders.

ARM II: Patients receive a reminder email survey every 2 weeks for 1 year after completing radiation.

ARM III: Patients receive a reminder email survey as in Arm I and 4 additional phone calls at 4-8 weeks, 3-5 months, 7-8 months, and 10-11 months during their first year of follow-up.

After completion of study, patients are followed up at 10-14 weeks, 5-7 months, 8-10 months, 11-13 months, 15-17 months, 19-21 months, and 23-25 months post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with gynecologic cancer who are undergoing vaginal brachytherapy as part of their treatment
* Patients cannot have previously received pelvic external beam radiation or brachytherapy. Patients may be enrolled while undergoing vaginal brachytherapy radiation treatment.
* Patients should have a life expectancy of at least 1 year
* No Eastern Cooperative Oncology Group (ECOG) or Karnofsky performance status requirements
* No organ and marrow function requirements
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have received prior pelvic external beam radiation or brachytherapy will be excluded
* No restrictions regarding use of other investigational agents
* No exclusion requirements due to co-morbid disease or intercurrent illness
* No investigational agent, so no exclusion requirements regarding history of allergic reactions attributed to compounds of similar chemical or biologic composition to investigational agent or device
* No exclusion criteria relating to concomitant medications
* No exclusion criteria for pregnant or nursing patients from participating in this study (Of note, pregnant patients will not be treated with vaginal brachytherapy, a requirement for enrolling on this study)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-09; Primary Completion 2019-01 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
Vaginal dilator adherence, measured by the average number of times per week patient uses a form of vaginal dilation | Up to 25 months after completing radiation
  The vaginal dilator adherence measurements will analyzed in repeated measures model with treatment as a fixed effect and time as a within subject effect. The overall mean of vaginal dilator adherence among the 3 groups will also be measured and compared. The interaction between treatment and time will also be tested to see if the behavior over time is different depending on which treatment arm the patient is in.

SECONDARY OUTCOMES:
Vaginal canal length | Up to 25 months after completing radiation
  The vaginal canal length will be measured using an extra small dilator and it will be calculated in centimeters. The vaginal canal length measurements will be analyzed in a repeated measures model with treatment as a fixed effect and time as a within subject effect. The interaction between treatment and time will also be tested to see if the behavior over time is different depending on which treatment arm the patient is in.
Incidence of adverse events (AE), reported by type and grade using the Common Terminology Criteria for Adverse Events version 4.03 | Up to 30 days after the last dose of study treatment
  The adverse events will be tabulated by type and grade at each follow up. The total number of AE's as well as the number of AE's in each category: gynecologic, urinary and gastrointestinal will tabulated. The test of proportion will be done per category of AE. Since it is possible that the rates will be low, an exact test will be used to compare the rates.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Kidd, Principal Investigator — Stanford University Hospitals and Clinics
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States